CLINICAL TRIAL: NCT05398224
Title: Phase II Study of Zanubrutinib in Combination With Rituximab and Methotrexate, Followed by Zanubrutinib Maintenance in Patients With Secondary Central Nervous System Lymphoma (SCNSL)
Brief Title: R-MTX-zanbrutinib in Secondary CNS Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Jun Zhu, professor, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20210218
Record Dates: First submitted 2022-05-22; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Secondary Central Nervous System Lymphoma
MeSH Terms: interventions — zanubrutinib; Methotrexate; Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm: Zanubrutinib, high-dose methotrexate (HD-MTX), rituximab (Experimental): Zanubrutinib in combination with rituximab and methotrexate, followed by zanubrutinib maintenance in patients with secondary central nervous system lymphoma (SCNSL)
  Interventions: Drug: Zanubrutinib, high-dose methotrexate (HD-MTX), rituximab

INTERVENTIONS:
Drug: Zanubrutinib, high-dose methotrexate (HD-MTX), rituximab — Induction therapy: Zanubrutinib will be given as 160mg bid orally between days 1 and 14 of each 14-day cycle; rituximab will be given at 375mg/m2 intravenously on day 1 of each cycle; methotrexate at 3.5g/m2 for patients ≤65 or 1.5g/m2 for patients >65 (standard hydration/leucovorin support) will be given intravenously on day 2 of each 14-day cycle; for 6 cycles.
  Consolidation therapy: For patients ≤65, autologous hematopoietic stem cell transplantation (ASCT with a conditioning regimen of thiotepa/carmustine) will be given as consolidation treatment after induction therapy.
  Maintenance therapy:Drug: zanubrutinib. Zanubrutinib will be given as 160mg bid orally continuously until progression of the disease (PD), intolerable toxicity, death, or patient/investigator discretion.

SUMMARY:
Secondary central nervous system lymphoma (SCNSL) occurred in about 5% of patients with diffuse large B-cell lymphoma (DLBCL). The prognosis of SCNSL is very poor. A number of retrospective studies have shown that the median overall survival (mOS) since the diagnosis of CNSL is only 2.5-3.5 months, and the 2-year OS rate is only 20%. At present, there is no consensus on the treatment of SCNSL, and new therapeutic strategies are urgently needed. Zanubrutinib is a new second-generation BTK inhibitor, which has showed good efficacy and safety in a variety of B-NHL. Zanubrutinib has showed good blood-brain barrier permeability in preclinical studies. This study attempts to evaluate the efficacy and safety of zanubrutinib combined with rituximab and high-dose methotrexate in the treatment of SCNSL in patients with DLBCL.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18, and ≤75 years of age
* Histologically documented systemic diffuse large B-cell lymphoma(DLBCL)
* Central nervous system (CNS) relapse (meningeal or /and intraparenchymal) with or without systemic lymphoma manifestations
* All patients need to have received at least one and ≤4 lines of prior therapy systemic lymphoma directed therapy.
* ECOG performance score 0-3
* Participants must have adequate bone marrow and organ function shown by:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L, Hemoglobin (Hgb) ≥ 9 g/dL, Platelets ≥ 75 x 109/L(≥ 50 x 109/L if bone marrow involvement)
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times the upper limit of normal, total bilirubin ≤ 2 times the upper limit of normal
  * International Normalized Ratio (INR) ≤ 1.5 and PTT (aPTT) ≤ 1.5 times the upper limit of normal
  * serum creatinine (mg/dL)) ≤ 1.5 times the upper limit of normal ; calculated creatinine clearance(CrCl) ≥ 40ml/min using the Cockcroft-Gault equation
* Expected survival greater than 3 months
* Did not receive targeting agents within 10 days or receive chemortherapy, radiotherapy, or monoclonal antibody within 3 weeks
* Woman of reproductive potential must agree to use highly effective methods of birth control during the period of therapy and for 30 days after the last dose of the study drug. Men who are sexually active must agree to use highly effective contraception during the period of therapy and for 3 months after the last dose
* Ability of participants or Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Newly diagnosed DLBCL with CNS involvement
* Previous treatment with Bruton's Tyrosine Kinase (BTK) inhibitors
* Received targeting agents within 10 days or received chemortherapy, radiotherapy, or monoclonal antibody within 3 weeks
* Patient has significant abnormalities on screening electrocardiogram (EKG) and active and significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, hypertension, valvular disease, pericarditis, or myocardial infarction within 6 months of screening
* History of severe bleeding diseases
* Patient is using warfarin or any other Coumadin-derivative anticoagulant or vitamin K antagonists. Patients must be off warfarin-derivative anticoagulants for at least seven days prior to starting the study drug. Low molecular weight heparin is allowed. Patients with congenital bleeding diathesis are excluded
* Patient is taking a drug known to be a moderate and strong inhibitor or inducers of the P450 isoenzyme CYP3A. Participants must be off P450/CYP3A inhibitors and inducers for at least two weeks prior to starting the study drug
* Patient is known to have human immunodeficiency virus (HIV) infection
* Patient is known to have a history of active or chronic infection with hepatitis C virus (HCV) or hepatitis B virus (HBV) as determined by serologic tests
* Patient is known to have an uncontrolled active systemic infection
* Patients with serous cavity effustion
* Patient underwent major systemic surgery ≤ 4 weeks prior to starting the trial treatment or who has not recovered from the side effects of such surgery
* Women who are pregnant or nursing (lactating)
* The patient is unwell or unable to participate in all required study evaluations and procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-02-26 (Actual); Primary Completion 2024-02-26 (Estimated); Study Completion 2024-05-26 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 1-year
  Progression-free survival (PFS) is defined as the time from the date of treatment start to the date of the first documented PD or death due to any cause

SECONDARY OUTCOMES:
Overall response rate (ORR) | at the end of 6 cycles of induction therapy (each cycle is 14 days)
Complete response (CR) | at the end of 6 cycles of induction therapy
Partial response (PR) | at the end of 6 cycles of induction therapy (each cycle is 14 days)
Overall survival (OS) | 1-year
safety/tolerability by assessing the frequency and severity of adverse events | at the end of 6 cycles of induction therapy (each cycle is 14 days), 1 year and 2 year maintenance therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality, China